CLINICAL TRIAL: NCT06127030
Title: The Effectiveness of a Brief Behavioral Training for Teachers of Children With Behavioral Difficulties at School: a Randomized Controlled Trial.
Brief Title: Brief Behavioral Teacher Training for Behavioral Difficulties
Acronym: PAINT-T
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Accare (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: METc 2023/183; PPO-RF-34 (Other Grant/Funding Number: PVO Researchfonds)
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Behavioral Difficulties; Behavioral Problem of Child
Keywords: Behavioral teacher training; Brief teacher training; Individually-tailored; School-based support

STUDY DESIGN:
Intervention Model Description: To examine the research objectives, a randomized controlled trial with two arms will be used. Teachers will be randomly assigned (equal randomization) to (a) brief teacher training with practice as usual (PAU) or (b) PAU only
Masking Description: N/A The investigator will not perform any outcome assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Brief behavioral teacher training and optional practice as usual (Experimental): A brief, individualized, three-session teacher training that exists of two (bi)weekly individually tailored training sessions of 120 minutes, and a third session of 60 minutes. Teachers and children may receive practice as usual as well. The practice as usual may include any support or treatment as regularly provided by mental health care centers, schools, school collaborations and/or other organizations, except from pharmacological treatment for children's behavioral difficulties and/or behavioral teacher training/support. Practice as usual can also imply that there is no support or treatment.
  Interventions: Behavioral: Brief behavioral teacher training
- Practice as usual only (PAU) (Active Comparator): PAU may include any support or treatment as regularly provided by mental health care centers, schools, school collaborations and/or other organizations, except from pharmacological treatment for children's behavioral difficulties and/or behavioral teacher training/support. PAU can also imply that there is no support or treatment. There are no criteria for professionals providing PAU.
  Interventions: Behavioral: Practice as usual only (PAU)

INTERVENTIONS:
Behavioral: Brief behavioral teacher training — A brief behavioral teacher training program that combines individually-tailored stimulus control and contingency management techniques to treat children's behavioral difficulties in two (bi)weekly training sessions of two hours and a third session of one hour in which the training will be evaluated and maintenance training will be provided.
  Other Names: The PAINT-T program; Brief teacher training
  Arms: Brief behavioral teacher training and optional practice as usual
Behavioral: Practice as usual only (PAU) — PAU may include any support or treatment as regularly provided by mental health care centers, schools, school collaborations and/or other organizations, except from pharmacological treatment for children's behavioral difficulties and/or behavioral teacher training/support. PAU can also imply that there is no support or treatment.
  Other Names: PAU
  Arms: Practice as usual only (PAU)

SUMMARY:
The goal of this two-armed randomized controlled trial is to investigate the effectiveness of a new, individually tailored, brief behavioral training for teachers of children with behavioral difficulties at school.

The main questions the study aims to answer are:

* Does the brief teacher training reduce the severity of four daily rated target behaviors in specific classroom situations compared to practice as usual (PAU) on the short term?
* Does the brief teacher training program reduce the severity of the same four daily rated target behaviors in other classroom situations, behavioral difficulties of the child at school and at home, and the impairment of the child in the school situation and reduce the number of behavioral difficulties of the child at school judged as troublesome by the teacher, and improve the teacher-student relationship quality, teachers' sense of efficacy, and teachers' behavior management strategies compared to practice as usual (PAU) on the short term?
* Are short-term improvements maintained at 3 months follow-up?

Teachers will be randomly assigned (simple randomization) to (a) three sessions of brief teacher training with PAU, or (b) PAU only. The brief teacher training provides teachers with individually tailored stimulus control and contingency management techniques to treat children's behavioral difficulties in two (bi)weekly training sessions of two hours and a third session of one hour in which the training will be evaluated and maintenance training will be provided. PAU may include any support or treatment as regularly provided by mental health care centers, schools, school collaborations and/or other organizations, except from pharmacological treatment for children's behavioral difficulties and/or behavioral teacher training/support. PAU can also imply that there is no support or treatment.

DETAILED DESCRIPTION:
INTRODUCTION AND RATIONALE

Behavioral difficulties, such as inattentive, impulsive, hyperactive, oppositional and/or aggressive behaviors, are highly prevalent in children and adolescents and one of the most common reasons for referral to mental health care. When left untreated, problems may exacerbate, grow into disorders and put children at risk of subsequent adverse outcomes, such as school dropout, delinquency, substance use, and/or depression. Ideally, treatment should prevent the escalation of problems, reduce the need for long and intensive treatments (including antipsychotics or other medication), and lower societal costs.

Behavioral teacher training is a promising intervention to treat children's behavioral difficulties at school. In the Netherlands, there are currently no brief and individual teacher training interventions available for this group of children. Existing programs are either self-help interventions, long programs that are not tailored to the individual teacher's and child's needs, or programs that focus on peer-support. There is thus an urgent need for a brief, accessible, and individually tailored teacher training programs.

To address this need, the Investigators will evaluate a brief, individually-tailored behavioral teacher training program based on effective training elements identified in our earlier work. Our previous project showed that effects of a brief teacher training on behavioral difficulties were promising, while the dropout rates of teachers were low. Teachers were particularly positive about the short time span of the training and the program's focus on tailoring program content to the individual problems that teachers and/or the child experience.

OBJECTIVES

Primary objective:

• To examine the short term effectiveness of a brief, individually-tailored, behavioral teacher training program on the severity of four daily rated target behaviors in specific classroom situations.

Secondary objectives:

* To examine the short term effectiveness of the teacher training on secondary outcome measures: the severity of the same four daily rated target behaviors in other classroom situations, behavioral difficulties of the child at school and at home, the number of behavioral difficulties of the child at school judged as troublesome by the teacher, and the impairment of the child in the school situation, the teacher-student relationship quality, teachers' sense of efficacy, and teachers' behavior management strategies.
* To examine the longer term effectiveness of the teacher training on primary and secondary outcomes.

STUDY DESIGN

The investigators will conduct a two-armed randomized controlled trial. Teachers will be randomly assigned (simple randomization) to (a) three sessions of brief teacher training with practice as usual (PAU), or (b) PAU only. Randomization will be done by a masked research assistant, who is not involved in the study, using a computer-generated randomized list.

The investigators will embed the trial in Dutch routine mental health care and Dutch school collaborations. Several school collaborations and at least two mental health care centers within the Netherlands will take part in the study.

In the intervention condition, primary and secondary outcome measures will be assessed before randomization (T0), one week after completion of the training (T1), and three months after T1 (T2). In the PAU condition primary and secondary outcome measures will be assessed before randomization (T0) and 8 weeks after T0 (T1). T2 does not apply for the PAU condition, as the brief teacher training can be provided in the PAU condition after T1 if needed. If T1 falls into a school vacation period, the measurement will be conducted during the first week following the school vacation.

TIME FRAME

November 2023: start recruitment, screening and inclusion of teachers and children, start running interventions.

November 2023-July 2025: ongoing contacts with participating mental health care organizations and school collaborations; recruitment, screening, and inclusion of teachers and children; run interventions and conduct measurements; supervision of therapists; fidelity checks; other project management activities.

July 2025-February 2028: data-checks and analysis, dissemination of results.

STUDY POPULATION

Participants will be Dutch elementary school teachers of children who display disruptive behaviors in the classroom in grade 1 to grade 8. The teachers work in a regular elementary school, a special elementary school or a special education school. The teachers (1) have been seeking help at school for handling the disruptive behavior of the child or (2) have a child in their classroom whose caretakers sought help at a mental health care institution for the disruptive behaviors of their child displayed at school. To enhance the generalizability of the results, the investigators aim to include a diverse sample of the Dutch population of children with disruptive behaviors, thus, from a broad age range (4-13 years), of both sexes, and all cultural and socioeconomic backgrounds

SAMPLE SIZE ASSESSMENT

In our prior randomized controlled study (with highly experienced therapists and no active interventions in the control group) the investigators found large short term effects on daily ratings of behavioral difficulties in the intervention group compared to waitlist (range of Cohen's d from .86 to .98;). For the current study the investigators estimated the short term effect of the brief teacher training as compared to PAU on our primary outcome measure to be at least small to medium (d = .35), as less experienced therapists will provide the training and children in both conditions can receive active interventions or support.

The investigators performed a power analysis (based on one primary outcome) using G*Power software. Based on the effect size of d = .35, two groups and two repeated measures, with r = .60 between-measurement relation, a power of .80 and alpha = .05, the investigators will need 27 participants per group, resulting in a total of 54 participants. The investigators increased the sample size by 10% as the investigators will have nested data resulting in 30 participants per group, leading to a total of 60 participants.

TREATMENT OF SUBJECTS

Brief teacher training The brief teacher training consists of three sessions. The first two sessions will both take 120 minutes and the third session will take one hour. These three sessions will be spread over a maximum of six weeks. In between sessions, teachers are asked to read some materials and execute the plan as made during the session.

The teacher training program uses the behavioral techniques that were identified as effective for behavioral difficulties in a microtrial of our group and in the broader literature. The program combines stimulus control and contingency management techniques that, separately, reduced behaviors difficulties in the previous microtrial.

In the screening phase, the teacher indicates which four, daily occurring, target behaviors in which specific situations they prefer to address in the training. These behaviors and situations will be sent to the trainer.

The program consists of four steps. First, psycho-education will be provided on executive function problems and motivational issues that may occur in children with behavioral difficulties. Second, using functional analyses, the trainer and teacher will decide which of the available techniques are most tailored to the first target behavior in a specific situation that individual teachers experience with their student. Third, the trainer and teacher make an action plan for the target behavior in the specific situations in which these techniques are included and explained to the teacher. Fourth, the action plan will be practiced using role play and the teacher is instructed to implement this plan as soon as possible in the classroom. In the second session, the steps will be repeated for a second problem behavior. In the third session, trainer and teacher evaluate both plans and discuss how to maintain and generalize the behavioral techniques that proved to work.

Trainers who provide the brief teacher training will be psychologists with a master's degree in psychology or educational science, higher professional education level mental health care professionals with postmaster cognitive behavioral training, or other mental health care professionals from schools who (1) have experience in supporting teachers and (2) have knowledge about behavioral therapy and psychopathology, as demonstrated by a completed higher professional education course including (or in addition) at least 150 hours of education on behavioral therapy and psychopathology.

The trainers need to participate in a one-day training provided by two experts in behavioral parent- and teacher training for which they are asked to read the materials carefully and need to submit a video in which they demonstrate certain aspects of the training. They will receive feedback from the experts or researchers on this video.

Practice as usual PAU may include any support or treatment as regularly provided by mental health care centers, schools, school collaborations and/or other organizations, except from pharmacological treatment for children's behavioral difficulties and/or behavioral teacher training/support. PAU can also imply that there is no support or treatment. There are no criteria for professionals providing PAU.

METHODS

Demographic information about the child and caregivers will be collected with a self-composed questionnaire (reported by caregivers) with questions about age and gender of the child and caregivers, educational background of the caregivers, and (possible) mental health disorders of the child. Also the teacher answers a self-composed questionnaire with questions about their age, gender, and educational background.

MODERATORS

As candidate moderators of treatment effects, the investigators will investigate:

* Class size;
* Treatment expectancy of the teacher, as measured with the Dutch translation of the Credibility and expectancy-scale of the teacher-rated Credibility and Expectancy Questionnaire (CEQ);
* Parent-reported child reward responsivity and punishment sensitivity, as measured with the Reward Responsiveness Scale and the Punishment Sensitivity Schale of the Sensitivity to Punishment and Sensitivity to Reward Questionnaire for Children (SPSRQ-C);
* Differential susceptibility, as measured with the Dutch translation of the caregiver-rated Highly Sensitive Child scale (HSC);
* Emotion regulation, as measured with the emotion regulation subscale of the Behavior Rating Inventory of Executive Function (BRIEF-2);
* Severity of behavioral difficulties of the child in the classroom at T0 (Intensity scale of the Dutch translation of the Sutter-Eyberg Student Behavior Inventory-Revised; SESBI-R);
* Quality of the teacher-student relationship (TSRS) at T0;
* Teacher-reported frequency of the use of supportive and non-supportive management strategies (TSQ) at T0.

STUDY PROCEDURES

Teachers will be recruited through:

(1) School collaborations, where teachers seek help for behavioral difficulties of one of their students; (2) Mental healthcare centers, where the child's caregiver(s) and/or the involved clinicians may indicate that help for behavioral difficulties of the concerning child is needed at school.

1. Recruitment through school collaborations:

   Healthcare professionals who work in schools will inform teachers who are seeking help for behavioral difficulties of a child about the study. If a teacher is interested in participating in the study, the healthcare professional or the teacher gets into contact with the caregiver(s) of the child and inform the teacher about the study. Caregivers may include parents with parental rights or legal guardians of the child. Caregivers and teachers who are interested in participating in the study need to give consent to share their contact information with the researcher through the healthcare professional from the school. The researchers will use this contact information to further inform teachers and caregivers about the study. If a teacher wants to participate, and caregivers also agree, they are both asked to provide informed consent. Both caregivers (if present) of the child have to provide consent. If the child is 12 years old or older, the child also needs to give informed consent. By default teachers, caregivers, and children 12 years or older have at least 14 days to decide upon participation and ask the researchers any questions.
2. Recruitment through mental healthcare centers:

Clinicians at the participating mental healthcare centers, who are involved in the treatment of a child who displays behavioral difficulties at school, will inform the caregiver(s) of the child about the study. If the caregivers are interested in the participation of the teacher of their child in the study, the clinician or caregivers then gets into contact with the teacher and informs him or her about the study. Caregivers and teachers who are interested can give consent to share their contact information with the researcher through the clinician. The researchers will use this contact information to further inform teachers and caregivers about the study. If teachers want to participate, and the caregivers also agree, they are both asked to provide informed consent. Both caregivers (if present) of the child are asked to provide consent. If the child is 12 years old or older, the child will also be asked to give informed consent. By default, teachers, caregivers, and children 12 years or older have at least 14 days to decide upon participation and ask the researchers any questions.

For teachers, completing the questionnaires at T1 and T2 will take a maximum of 30 minutes. At T0, additional questionnaires will be administered for intended moderation analyses (extra 10 minutes, maximum 40 minutes in total). The phone calls to the teacher will take two to three minutes each, on four consecutive days per measurement occasion.

For caregivers, the questionnaires at T1 and T2 will take a maximum of 15 minutes. At T0, additional questionnaires will be administered for intended moderation analyses (extra 10 minutes, maximum 25 minutes in total).

STATISTICAL ANALYSIS

PRIMARY AND SECONDARY STUDY PARAMETERS

Data will be analyzed on an intention-to-treat basis. Differences in demographic variables between the study-arms will be analyzed with ANOVA's (continuous variables) or chi-squared tests (categorical variables). To examine the effects of the intervention on the primary and secondary outcomes the investigators will conduct multilevel analyses (mixed modeling). Mixed model analyses take missing data into account (Twisk et al., 2013). The investigators test a three-level multilevel model: outcomes (level 1), nested within children (level 2), nested within trainers (level 3). For trainers (level 3), the investigators will test whether including the level will result in a better model fit. If not, the level will not be taken into account.

MODERATORS

To assess the influence of candidate moderating variables on treatment effects, the investigators will include these variables as interaction effects in the multilevel analysis.

ETHICAL CONSIDERATIONS

The risk of any physical or mental harm caused by the study is very low and not to be expected higher than what may be expected in the daily practice of the teacher or in the daily school life of students. The investigators will exclusively use conventional methods and interventions. The study is embedded in mental healthcare settings and school collaborations.

The children will not directly be involved in the study. They will not be present during the brief teacher training sessions and all measures will be parent- or teacher-reported measures.

Teachers, caregivers and/or children 12 years old or older can decide to leave the study at any time for any reason if they wish to do so without any consequences.

To debrief teachers, caregivers, and children 12 years or older who wish to learn about the results of the study can request this information from the researchers after the study is finished. This concerns only information on group level. The investigators will inform teachers and caregivers about the possibility to ask for this information in the information letter.

ADMINISTRATIVE ASPECTS, MONITORING AND PUBLICATION

HANDLING AND STORAGE OF DATA AND DOCUMENTS

Digital data, both raw and processed/analyzed data will be stored at a study specific highly secured folder within the Accare network. This study specific folder can only be accessed by researchers involved in this study.

All phone and questionnaire data and processed audio files (which are use to score treatment integrity, see below for more details) will be stored in one, pseudonymized file, that is accompanied by a 'readme' text file that contains a code book explaining the meaning of all variables. The file contains separate pages ('tabs') for all different outcome variables at all different timepoints. A separate logbook-file will be created documenting all decisions that will be made during the process from raw to published data. Old versions of all these documents will be stored, document names will contain their date to ensure version control.

Management of the data and access permissions are with the principal investigators of the research project.

Access permissions are controlled by the research project's principal investigators. Raw data containing identifiable information such as the separate log containing patient identification number and study code will be kept strictly separate from the processed data (in a separate folder) and can only be accessed by the supervisors, research assistants and PhD student. The processed, pseudonymized data will be available for fellow researchers and made available (restricted access) for re-use. Requests for re-use of data after the completion of the research project will be evaluated by principal investigators BvdH, TD, and ML who will check whether the research question falls within the scope of the informed consent.

After the research project has been completed (i.e., after data collection, data analysis and publishing of articles) all the anonymized (i.e., the link with identifiable information will be deleted) digital data will be transferred to a study specific folder for long-term storage within the Accare network. The folder can only be accessed by the principal investigators and by authorized personnel after approval of the Principal Investigators. This data storage environment allows for careful access management and is only accessible with username and password. Data storage is backed-up automatically daily.

All the research data will be stored for 15 years after the data collection has been completed (i.e. last research assessment for the last patient has been performed). Raw audio-files, that may contain personal information, will be stored for 15 years in an encrypted folder.

MONITORING AND QUALITY ASSURANCE

Not applicable.

INERVENTION INTEGRITY

Intervention integrity will be assessed using an adapted version of the procedures of Abikoff. All intervention sessions will be audiotaped. For every trainer, the first session will be checked and they will receive feedback on intervention integrity and fidelity by a cognitive behavioral therapist with extensive experience in behavioral teacher training.

Further, audiotapes of a subset of randomly selected sessions will be scored on intervention integrity and fidelity during the study by independent evaluators. In addition, after each session, the trainers have to complete a fidelity checklist in which they will be asked which topics were covered.

ELIGIBILITY:
Inclusion criteria for the teachers will be:

1. The teacher works in regular elementary education, special elementary education or special education (in Dutch: cluster 4);
2. The teacher indicates that the child displays at least four behavioral difficulties in the classroom on a daily basis that the teacher wants to target in the training (using a list of target disruptive behaviors (Hornstra et al., 2021; Van den Hoofdakker et al., 2007)).

Exclusion criterion for the teachers will be:

1. The teacher has received behavioral training or behavioral support aimed at remediating behavioral difficulties of the concerned child within the past year;
2. The teacher already participates in the study with another child.

Exclusion criteria for the children will be:

1. The child has a diagnosis of autism spectrum disorder (as reported by parents, we will not perform any measures to assess autism spectrum disorder);
2. The child currently receives pharmacological treatment for behavioral difficulties (e.g., methylphenidate).

Ages: 4 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2025-07-04 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Severity of four daily rated target behaviors in specific classroom situations | Before randomization (T0), one week after the brief training (experimental arm)/eight weeks after T0 (control arm) (T1), three months after T1 (T2, experimental arm only)
  The primary outcome measure will be the severity of teacher-rated daily measured target behaviors in specific classroom situations. Teachers select four daily occurring behavioral difficulties of the child in the classroom (i.e., target behaviors of the intervention) and the specific situations. Target behaviors will be selected from an adapted version of a list (Hornstra et al., 2021; Van den Hoofdakker et al., 2007), with teachers indicating daily occurrence (yes/no) and rating severity on a 5-point Likert scale (1=not severe to 5=extremely severe). Specific classroom situations will be selected from the School Situation questionnaire (SSQ-R; DuPaul & Barkley, 1992). Severity of the target behaviors in these specific situations will be measured with brief daily phone calls to teachers on four consecutive school days, by the researchers. Teachers report whether the four selected target behaviors occurred (yes/no) and rate their severity on a 5-point scale.

SECONDARY OUTCOMES:
Severity of daily the same four daily rated target behaviors in other classroom situations than the specified situation which is used as primary outcome (see primary outcome measure for details on administration) | Before randomization (T0), one week after the brief training (experimental arm)/eight weeks after T0 (control arm) (T1), three months after T1 (T2, experimental arm only)
  To investigate whether the four target behaviors improve in other situations, we will ask teachers during the daily phone calls if these behaviors occurred in any of the other situations of the SSQ-R (DuPaul & Barkley, 1992) (yes/no) in the last day the teacher had contact with the child. Items scored as 'yes' will be rated on a 5-point Likert scale ranging from 1 (not severe) to 5 (extremely severe).
Teacher-reported severity of behavioral difficulties of the child in the classroom | Before randomization (T0), one week after the brief training (experimental arm)/eight weeks after T0 (control arm) (T1), three months after T1 (T2, experimental arm only)
  Severity of children's behavioral difficulties in the classroom will be measured with the Intensity scale of the Dutch version of the Sutter-Eyberg Student Behavior Inventory-Revised (SESBI-R; Eyberg & Pincus, 1999). On 38 items, teachers have to rate the frequency of the child's behavioral difficulties on a 7-point Likert scale, ranging from 1 (never) to 7 (always).
Teacher-reported number of child behavioral difficulties in the classroom that the teacher considers troublesome | Before randomization (T0), one week after the brief training (experimental arm)/eight weeks after T0 (control arm) (T1), three months after T1 (T2, experimental arm only)
  The number of children's behavioral difficulties in the classroom which the teacher considers troublesome will be measured with the Problem subscale of the Dutch version of the Sutter-Eyberg Student Behavior Inventory-Revised (SESBI-R; (Eyberg & Pincus, 1999)). On 38 items, teachers have to indicate if the behavioral difficulties are problem for them by answering yes (0) or no (1).
Teacher-reported child impairment at school associated with behavioral difficulties | Before randomization (T0), one week after the brief training (experimental arm)/eight weeks after T0 (control arm) (T1), three months after T1 (T2, experimental arm only)
  Children's impairment associated with behavioral difficulties at school will be measured with a slightly adapted (i.e., we asked the teachers to specifically link the impairment to the behavioral difficulties) version of the Dutch version of the impairment rating scale - Teacher (IRS-T; Fabiano et al., 2006). On 6 items, teachers have to rate the impairment of the child on a 7-point Likert scale, ranging from no problem (0) to extreme problem (6).
Teacher-reported quality of the teacher-student relationship | Before randomization (T0), one week after the brief training (experimental arm)/eight weeks after T0 (control arm) (T1), three months after T1 (T2, experimental arm only)].
  The quality of the teacher-student relation will be measured with the Student-Teacher Relationship Scale - short version (STRS; Koomen et al., 2012; Pianta, 1992). On 15 items, teachers have to rate their relationship with their student on a 5-point Likert scale, ranging from 1 (definitely does not apply) to 5 (definitely applies).
Teacher's sense of self-efficacy | Before randomization (T0), one week after the brief training (experimental arm)/eight weeks after T0 (control arm) (T1), three months after T1 (T2, experimental arm only)
  Teachers' sense of self-efficacy will be measured with the short version of the Teachers' Sense of Efficacy Scale (TSES; Tschannen-Moran & Hoy, 2001). On 12 items, teachers have to rate their sense of self-efficacy on a 9-point Likert scale, ranging from 1 (I can do nothing) to 9 (I can do a great deal).
Teacher-reported frequency of supportive and non-supportive management strategies | Before randomization (T0), one week after the brief training (experimental arm)/eight weeks after T0 (control arm) (T1), three months after T1 (T2, experimental arm only
  Teacher behavior will be assessed with two subscales (frequency of Positive Management Strategies and frequency of Inappropriate Management Strategies, respectively) of the Teacher Strategy Questionnaire (TSQ; Webster-Stratton et al., 2001). The Positive Management Strategies subscale contains 18 items, the Inappropriate Management Strategies contains 9 items. Items are answered on a 5-point Likert scale, ranging from rarely/ never (1) to very often (5). We will only use the items focused on the frequency of the strategy use.
Caregiver-reported severity of child behavioral difficulties at home | Before randomization (T0), one week after the brief training (experimental arm)/eight weeks after T0 (control arm) (T1), three months after T1 (T2, experimental arm only)
  Severity of children's behavior difficulties at home will be measured with the 36-item Intensity scale of the Dutch version of the Eyberg Child Behavior Inventory (ECBI-I; Eyberg & Pincus, 1999), on which the caregiver rates the frequency of specific behavioral difficulties on a 7-point Likert scale from 1 (never) to 7 (always).

OTHER OUTCOMES:
Teacher/school-reported history of mental healthcare/support. | Before randomization (T0)
  A self-developed questionnaire will be used to measure the history of mental healthcare/support for the behavioral difficulties of the considering child (including teacher support/training and programs for all children in the classroom)
Teacher/school-reported use of mental health care or support for behavioral difficulties of the child in the classroom | One week after the brief training (experimental arm)/eight weeks after T0 (control arm) (T1)
  A self-developed questionnaire will be used to assess the use of mental health care or support for of the child in the classroom (including teacher support/training and programs for all children in the classroom) in the period between T0 and T1.
Caregiver-reported history of mental healthcare/support | Before randomization (T0)
  A self-developed questionnaire will be used to measure the history of mental healthcare/support (except care/support provided at school) for the behavioral difficulties of the child.
Caregiver-reported use of mental health care for behavioral difficulties of the child at home. | One week after the brief training (experimental arm)/eight weeks after T0 (control arm) (T1).
  A self-developed questionnaire will be used to assess the use of mental health care/support (except health care/support provided at school) for behavioral difficulties displayed by the child in the period between T0 and T1.
Teachers satisfaction with the teacher training | One week after the brief training (experimental group only) (T1).
  Teachers' satisfaction with the brief training will be measured with a self-developed satisfaction questionnaire, which is based on questions of the Parent Satisfaction Questionnaire (Bearss et al., 2013), the Therapy Attitude Inventory (Eyberg & Johnson, 1974), and the satisfaction questionnaire that was used in Breider et al. (2018). Teachers have to answer 15 questions about their satisfaction with the training on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree) and give the brief teacher training a grade between 1 (very bad) and 10 (excellent).
Adverse reactions to the teacher training | One week after the brief training (experimental arm)/eight weeks after T0 (control arm) (T1), and at T2.
  Adverse effects of the teacher training will be measured with a self-developed adverse effects questionnaire filled out by the teacher. On six items teachers indicate possible adverse reactions.
Teacher/school-reported use of mental health care or support for behavioral difficulties of the child in the classroom | Three months after T1 (T2)
  A self-developed questionnaire will be used to assess the use of mental health care or support for of the child in the classroom (including teacher support/training and programs for all children in the classroom) in the period between T1 and T2.
Caregiver-reported use of mental health care for behavioral difficulties of the child at home | Three months after T1 (T2)
  A self-developed questionnaire will be used to assess the use of mental health care/support (except health care/support provided at school) for behavioral difficulties displayed by the child in the period between T1 and T2.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara van den Hoofdakker, Prof. dr., Principal Investigator — Accare child study centre; University Medical Center Groningen; Marjolein Luman, Dr., Principal Investigator — Free university of Amsterdam; Saskia van der Oord, Prof. dr., Principal Investigator — KU Leuven; Tycho Dekkers, Dr, Principal Investigator — Accare child study centre; University Medical Center Groningen
Locations (1):
- Accare Child Study Center, Groningen, Provincie Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abikoff HB, Thompson M, Laver-Bradbury C, Long N, Forehand RL, Miller Brotman L, Klein RG, Reiss P, Huo L, Sonuga-Barke E. Parent training for preschool ADHD: a randomized controlled trial of specialized and generic programs. J Child Psychol Psychiatry. 2015 Jun;56(6):618-31. doi: 10.1111/jcpp.12346. Epub 2014 Oct 16. PMID 25318650
- [Background] Abikoff H, Gallagher R, Wells KC, Murray DW, Huang L, Lu F, Petkova E. Remediating organizational functioning in children with ADHD: immediate and long-term effects from a randomized controlled trial. J Consult Clin Psychol. 2013 Feb;81(1):113-28. doi: 10.1037/a0029648. Epub 2012 Aug 13. PMID 22889336
- [Background] Bearss K, Lecavalier L, Minshawi N, Johnson C, Smith T, Handen B, Sukhodolsky D, Aman M, Swiezy N, Butter E, Scahill L. Toward an exportable parent training program for disruptive behaviors in autism spectrum disorders. Neuropsychiatry (London). 2013 Apr;3(2):169-180. doi: 10.2217/npy.13.14. PMID 23772233
- [Background] Breider S, de Bildt A, Nauta MH, Hoekstra PJ, van den Hoofdakker BJ. Self-directed or therapist-led parent training for children with attention deficit hyperactivity disorder? A randomized controlled non-inferiority pilot trial. Internet Interv. 2019 Aug 8;18:100262. doi: 10.1016/j.invent.2019.100262. eCollection 2019 Dec. PMID 31890615
- [Background] Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry. 2000 Jun;31(2):73-86. doi: 10.1016/s0005-7916(00)00012-4. PMID 11132119
- [Background] Drummond et al., (2015). Methods for the economic evaluation of health care programs (Fourth edition). Oxford University Press.
- [Background] DuPaul, G. J., & Barkley, R. A. (1992). Situational Variability of Attention Problems: Psychometric Properties of the Revised Home and School Situations Questionnaires. Journal of Clinical Child Psychology, 21(2), 178-188. https://doi.org/10.1207/S15374424JCCP2102_10
- [Background] Eyberg SM, Johnson SM. Multiple assessment of behavior modification with families: effects of contingency contracting and order of treated problems. J Consult Clin Psychol. 1974 Aug;42(4):594-606. doi: 10.1037/h0036723. No abstract available. PMID 4847264
- [Background] Eyberg, S. M., & Pincus, D. (1999). Eyberg Child Behavior Inventory and Sutter-Eyberg Student Behavior Inventory: Professional manual. Psychological Assessment Resources.
- [Background] Fabiano GA, Pelham WE Jr, Waschbusch DA, Gnagy EM, Lahey BB, Chronis AM, Onyango AN, Kipp H, Lopez-Williams A, Burrows-Maclean L. A practical measure of impairment: psychometric properties of the impairment rating scale in samples of children with attention deficit hyperactivity disorder and two school-based samples. J Clin Child Adolesc Psychol. 2006 Sep;35(3):369-85. doi: 10.1207/s15374424jccp3503_3. PMID 16836475
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Franke N, Keown LJ, Sanders MR. An RCT of an Online Parenting Program for Parents of Preschool-Aged Children With ADHD Symptoms. J Atten Disord. 2020 Oct;24(12):1716-1726. doi: 10.1177/1087054716667598. Epub 2016 Sep 8. PMID 27609783
- [Background] Hornstra R, van der Oord S, Staff AI, Hoekstra PJ, Oosterlaan J, van der Veen-Mulders L, Luman M, van den Hoofdakker BJ. Which Techniques Work in Behavioral Parent Training for Children with ADHD? A Randomized Controlled Microtrial. J Clin Child Adolesc Psychol. 2021 Nov-Dec;50(6):888-903. doi: 10.1080/15374416.2021.1955368. Epub 2021 Aug 23. PMID 34424102
- [Background] Kaminski JW, Valle LA, Filene JH, Boyle CL. A meta-analytic review of components associated with parent training program effectiveness. J Abnorm Child Psychol. 2008 May;36(4):567-89. doi: 10.1007/s10802-007-9201-9. Epub 2008 Jan 19. PMID 18205039
- [Background] Koomen HM, Verschueren K, van Schooten E, Jak S, Pianta RC. Validating the Student-Teacher Relationship Scale: testing factor structure and measurement invariance across child gender and age in a Dutch sample. J Sch Psychol. 2012 Apr;50(2):215-34. doi: 10.1016/j.jsp.2011.09.001. Epub 2011 Oct 5. PMID 22386121
- [Background] Leijten P, Gardner F, Melendez-Torres GJ, van Aar J, Hutchings J, Schulz S, Knerr W, Overbeek G. Meta-Analyses: Key Parenting Program Components for Disruptive Child Behavior. J Am Acad Child Adolesc Psychiatry. 2019 Feb;58(2):180-190. doi: 10.1016/j.jaac.2018.07.900. Epub 2018 Nov 26. PMID 30738545
- [Background] Leijten P, Melendez-Torres GJ, Gardner F. Research Review: The most effective parenting program content for disruptive child behavior - a network meta-analysis. J Child Psychol Psychiatry. 2022 Feb;63(2):132-142. doi: 10.1111/jcpp.13483. Epub 2021 Jul 9. PMID 34240409
- [Background] Luman M, van Meel CS, Oosterlaan J, Geurts HM. Reward and punishment sensitivity in children with ADHD: validating the Sensitivity to Punishment and Sensitivity to Reward Questionnaire for children (SPSRQ-C). J Abnorm Child Psychol. 2012 Jan;40(1):145-57. doi: 10.1007/s10802-011-9547-x. PMID 21789519
- [Background] Pianta, R. C. (1992). Student-teacher relationship scale - Short form. Psychological Assessment Resources.
- [Background] Pluess M, Assary E, Lionetti F, Lester KJ, Krapohl E, Aron EN, Aron A. Environmental sensitivity in children: Development of the Highly Sensitive Child Scale and identification of sensitivity groups. Dev Psychol. 2018 Jan;54(1):51-70. doi: 10.1037/dev0000406. Epub 2017 Sep 21. PMID 28933890
- [Background] Reef J, Diamantopoulou S, van Meurs I, Verhulst FC, van der Ende J. Developmental trajectories of child to adolescent externalizing behavior and adult DSM-IV disorder: results of a 24-year longitudinal study. Soc Psychiatry Psychiatr Epidemiol. 2011 Dec;46(12):1233-41. doi: 10.1007/s00127-010-0297-9. Epub 2010 Oct 10. PMID 20936464
- [Background] Slagt M, Dubas JS, van Aken MAG, Ellis BJ, Dekovic M. Sensory processing sensitivity as a marker of differential susceptibility to parenting. Dev Psychol. 2018 Mar;54(3):543-558. doi: 10.1037/dev0000431. Epub 2017 Nov 20. PMID 29154642
- [Background] Sperati A, Spinelli M, Fasolo M, Pastore M, Pluess M, Lionetti F. Investigating sensitivity through the lens of parents: validation of the parent-report version of the Highly Sensitive Child scale. Dev Psychopathol. 2024 Feb;36(1):415-428. doi: 10.1017/S0954579422001298. Epub 2022 Dec 12. PMID 36503569
- [Background] Staff AI, van den Hoofdakker BJ, van der Oord S, Hornstra R, Hoekstra PJ, Twisk JWR, Oosterlaan J, Luman M. Effectiveness of Specific Techniques in Behavioral Teacher Training for Childhood ADHD: A Randomized Controlled Microtrial. J Clin Child Adolesc Psychol. 2021 Nov-Dec;50(6):763-779. doi: 10.1080/15374416.2020.1846542. Epub 2021 Jan 20. PMID 33471581
- [Background] Tschannen-Moran, M., & Hoy, A. W. (2001). Teacher efficacy: capturing an elusive construct. Teaching and Teacher Education, 17(7), 783-805. https://doi.org/10.1016/S0742-051X(01)00036-1
- [Background] Twisk J, de Boer M, de Vente W, Heymans M. Multiple imputation of missing values was not necessary before performing a longitudinal mixed-model analysis. J Clin Epidemiol. 2013 Sep;66(9):1022-8. doi: 10.1016/j.jclinepi.2013.03.017. Epub 2013 Jun 21. PMID 23790725
- [Background] van den Hoofdakker BJ, van der Veen-Mulders L, Sytema S, Emmelkamp PMG, Minderaa RB, Nauta MH. Effectiveness of behavioral parent training for children with ADHD in routine clinical practice: a randomized controlled study. J Am Acad Child Adolesc Psychiatry. 2007 Oct;46(10):1263-1271. doi: 10.1097/chi.0b013e3181354bc2. PMID 17885567
- [Background] Ward RJ, Bristow SJ, Kovshoff H, Cortese S, Kreppner J. The Effects of ADHD Teacher Training Programs on Teachers and Pupils: A Systematic Review and Meta-Analysis. J Atten Disord. 2022 Jan;26(2):225-244. doi: 10.1177/1087054720972801. Epub 2020 Dec 17. PMID 33331193
- [Background] Webster-Stratton C, Reid MJ, Hammond M. Preventing conduct problems, promoting social competence: a parent and teacher training partnership in head start. J Clin Child Psychol. 2001 Sep;30(3):283-302. doi: 10.1207/S15374424JCCP3003_2. PMID 11501247